CLINICAL TRIAL: NCT07278089
Title: Screening of Atrial Fibrillation/Arrhythmia Events in Patients With Abnormal Echocardiographic Parameters: The Randomized, Prospective SAFE-ECHO Study Design and Rationale
Brief Title: AF Screening in Patients With Abnormal Echocardiographic Parameters
Acronym: SAFE-ECHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tze-Fan Chao (Other Government)
Responsible Party: Sponsor-Investigator, Tze-Fan Chao, Doctor, Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-01-001BC; NSTC 113-2628-B-075 -002 -MY3 (Other: Ministry of Science and Technology, Taiwan)
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study arm (Active Comparator)
  Interventions: Diagnostic Test: study arm
- control arm (No Intervention)

INTERVENTIONS:
Diagnostic Test: study arm — Scheduled cardiac rhythm monitoring every 3 months using extended continuous ECG monitoring
  Arms: study arm

SUMMARY:
To evaluate the feasibility of specific echocardiographic parameters as criteria for AF screening and to determine the AF detection yield of scheduled extended ECG monitoring compared to contemporary care.

ELIGIBILITY:
Inclusion Criteria: patients who met any of the following criteria

1. LAE: defined as LAD ≥ 45 mm or LAVI > 34 ml/m2;
2. LVH: defined as LV septal or posterior wall thickness ≥ 15 mm;
3. E/e' > 14;
4. grade II or III diastolic dysfunction;
5. VHD;
6. HF: defined as LVEF < 40% or LVEF ≥40% with clinical presentation compatible with Framingham criteria, New York Heart Association functional classification II-IV, and N-terminal pro-B type natriuretic peptide (NT-proBNP) > 125 pg/ml.

Exclusion Criteria:

* Patients with a history of AF or atrial flutter, congenital heart disease, acute coronary syndrome undergoing urgent percutaneous coronary intervention within 3 months, uncontrolled hyperthyroidism, end-stage renal disease, unstable hemodynamic status or any known major comorbidities or medical conditions with expected life expectancy less than 1 year are excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
the detection of AF either by 12-lead ECG or any episodes of AF lasting ≥ 30 seconds by the single-lead ECG or 7-day continuous recording. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided